CLINICAL TRIAL: NCT02397681
Title: Autonomic Responses During the Valsalva Maneuver and Deep Breathing Test Depend on the Experimental Setup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Aalborg University (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AUTO-2015
Record Dates: First submitted 2015-02-11; First posted 2015-03-25 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Autonomic Nervous System Diseases
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Autonomic Function Testing

INTERVENTIONS:
Other: Autonomic Function Testing — Autonomic nervous system index assessed with Task Force Monitor (CNSystems Medizintechnik AG, Graz, Austria)

SUMMARY:
The purpose of this study is to determine the effects of procedural differences during the Valsalva maneuver and deep breathing test in autonomic nervous system testing.

ELIGIBILITY:
Inclusion Criteria:

* male
* ≥ 18 year
* normal ECG-12

Exclusion Criteria:

* any known disease
* smoking
* any intake of regular medicine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure changes to cardiovascular adrenergic activation | 3 hours
Heart rate changes to parasympathetic activation | 3 hours

SECONDARY OUTCOMES:
Expiratory pressure during the Valsalva maneuver | 3 hours
Expiratory duration during the Valsalva maneuver | 3 hours
Air volume exchanged per respiratory cycle during deep respiration | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Astrid J. Terkelsen, Principal Investigator — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark